CLINICAL TRIAL: NCT06075069
Title: Evaluation of the Effect of Prosthetic Management for Congenital Cleft Lip and Palate Infants on the Middle Ear Function: Clinical Trial
Brief Title: Evaluation of the Effect of Prosthetic Management for Congenital Cleft Lip and Palate Infants on the Middle Ear Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Kamel Salah, Assistant Lecturer of Prosthodontics, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #111
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Feeding appliance immediately after birth (Experimental)
  Interventions: Device: Feeding appliance
- Feeding appliance after 1-3 months (Experimental)
  Interventions: Device: Feeding appliance
- Feeding appliance after 4 -12 months (Experimental)
  Interventions: Device: Feeding appliance

INTERVENTIONS:
Device: Feeding appliance — A preliminary alginate impression was made using wax stock tray to get a preliminary cast and construct a self-cure acrylic custom-made tray. A Medium viscosity rubber base impression material was used for making final impression which in turn will be poured to obtain a master cast. On this master cast, a feeding appliance will be constructed. Readymade facebow with two straight side length of hard, rounded, of 2mm diameter, 15cm length Nickel-Chrome wire with omega loops (at the end of the wire) was used to form extra-oral wings to be used as a retentive aid to maintain the prosthesis in situ. The appliance was fabricated in clear acrylic resin then finished and polished. A small piece of cold cure acrylic resin was added and adapted to the omega loops and manipulated to follow the checks contour.

SUMMARY:
Aim of the study was to evaluate the effect of feeding appliance for congenital cleft lip and palate infants on the middle ear function

ELIGIBILITY:
Inclusion Criteria:

* Infants with bilateral cleft lip and palate.
* Centralized pre-maxilla that does not need active appliance.
* Normal inner ear and auditory nerve function.

Exclusion Criteria:

* Infant with unilateral cleft lip and palate or cleft palate only.
* Deviated pre-maxilla that needs active appliance.
* Congenital hearing problems or sensorineural hearing loss/

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Assessment of middle ear pressure | up to one year of age
  This was performed using Tympanometer that measures the air pressure in the middle ear to obtain Tympanogram which is a graphic representation of how the eardrum moves in response to the air pressure in the ear canal. Tympanometry was performed using a AT235 tympanometer with a 226-Hz probe frequency. It was calibrated to ANSI standards (American National Standards Institute,1987).
  The normal middle-ear pressure values for children are +50 daPa to -200 daPa.
Assessment of middle ear compliance | up to one year of age
  This was performed using Tympanometer.
  The patients' tympanometric results were classified into three types:
  * Type A: Static compliance greater than 0.1 ml and the point of greatest compliance is at approximately 0 daPa; the curve is shown by a large, inverted V. In a "type A" curve, the peak compliance occurs at or near atmospheric pressure indicating normal pressure within the middle ear.
  * Type B: The point of greatest compliance cannot be found, and the curve is shown by a flat curve (no peak). This is indicative of non-compressible fluid within the middle ear space (otitis media), tympanic membrane perforation, or debris within the external ear canal.
  * Type C: Static compliance greater than or equal to 0.2 ml, and the peak compliance is significantly below zero (usually less than -200), indicating negative pressure (sub-atmospheric) within the middle ear space.
  Type A tympanograms were classified as normal, but types B and C were considered abnormal
Assessment of hearing quality | up to one year of age
  Audiometric screening will be performed using Auditory brainstem response (ABR) conducted under natural sleep as far as possible. ABR can provide information about the softest level of sound the ear can hear. It is traditionally used to determine the degree of hearing loss in pediatrics.
  ABR test uses electrodes attached with adhesive to the baby's scalp. While the baby is sleeping, clicking sounds were made through headphones over the baby's ears. The test measures the brain's activity in response to the sounds.
  Hearing level thresholds as estimated by ABR are categorized as normal (25 - 35 dB nHL), mild (35 - 45 dB nHL), moderate (45 - 65 dB nHL), severe (65 - 90 dB nHL), and profound (90 dB nHL) hearing loss.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt